CLINICAL TRIAL: NCT02743468
Title: Cytochrome P450 Epoxygenase Pathway Regulation of Macrophage Function
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 160096; 16-E-0096
Record Dates: First submitted 2016-04-14; First posted 2016-04-19 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2025-06-02

CONDITIONS: Polymorphism; Lung Inflammation
Keywords: Bronchoscopy; Pollutants; Human Pulmonary Cells; Macrophage Function; Soluble Epoxide Hydrolase; Natural History
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Volunteers: Healthy Volunteers

SUMMARY:
Background:

Respiratory diseases affect more than 1 billion people worldwide. They are a growing public health concern. The lungs are constantly exposed to environmental factors such as dust, fumes, microbes, and pollutants. But much is still not known about how these pollutants lead to respiratory illnesses. Researchers want to collect samples from lungs and blood to see how genetics and environmental pollutants affect cellular responses or functioning.

Objectives:

To study how cytochrome P450 epoxygenase pathway enzymes affect macrophage function in the lungs and inflammatory responses.

Eligibility:

Adults ages 18 65 who can have a bronchoscopy.

Design:

All study visits will take place at the NIEHS Clinical Research Unit in Research Triangle Park, NC.

At study visit 1, participants will be screened with medical history and physical exam. They will have blood and urine tests. They will take tests that measure their lung function. They will answer questionnaires. Before the visit, they will be given a list of medicines they cannot take. They also must not have caffeine on the day of their visit. The visit will last about 3 hours.

At study visit 2, participants will give blood samples. They will undergo bronchoscopy. For this, they will get an intravenous line in a vein to get sedatives. Their airways will be numbed. Cells will be collected from their lungs. They will fast for 8 hours before the visit. They must have someone else drive them home from the visit. The visit will last about 3-4 hours.

Participants will get a follow-up phone call about 1 day after study visit 2.

DETAILED DESCRIPTION:
This is a prospective, cross-sectional study designed to provide a consistent method for obtaining biological samples and respiratory health-related information from participants for use in research that evaluates lung function (e.g., responses to environmental agents such as air pollution particles, engineered nanomaterials, or immune ligands; the role of genetics on cellular responses or functioning).

Study participants will be adult volunteers, ages 18-65 (inclusive), who meet eligibility criteria to undergo bronchoscopy. Potential participants will be prescreened and scheduled for a final eligibility visit that will include medical history review, vital signs, physical examination, blood draw, and pulmonary function tests. After eligibility is confirmed, the participant will be scheduled for biological sample collections, which will include a blood draw and bronchoscopy.

The objective of this protocol is to investigate the role of cytochrome P450 (CYP) epoxygenase pathway enzymes, including the soluble epoxide hydrolase (sEH; encoded by EPHX2) and CYP2J2 proteins, in macrophage function and inflammatory responses. The primary outcome measure will evaluate macrophage phagocytosis in an ex vivo assay, comparing groups of individuals with and without EPHX2 and CYP2J2 polymorphisms of interest. Secondary outcomes will include evaluations of ex vivo gene expression of inflammatory receptors and cytokines in stimulated macrophages (alveolar and peripheral blood monocyte-derived), assessment of the lower airway microbiome from bronchoalveolar lavage (BAL) fluid, and measurement of eicosanoids and cytokines in serum and BAL fluid.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Age 18 to 65 years, inclusive (males and females)
  2. Able to travel to the NIEHS CRU for required study visits
  3. Able to present a valid government-issued form of identification for entry to the NIEHS campus
  4. Able to fast for 8 hours prior to the visit where bronchoscopy occurs
  5. Has a responsible party who is willing and able to attend Visit 2 and drive the participant away from the CRU after completion of Visit 2, if the participant elects to undergo conscious sedation
  6. Genotype information available for relevant CYP2J2 and EPHX2 polymorphisms, which indicates:
* Wild type with respect to EPHX2 K55R, EPHX2 R287Q, and CYP2J2*7; or
* Homozygous for EPHX2 K55R (wild type for the other SNPs); or
* Homozygous for EPHX2 R287Q (wild type for the other SNPs); or
* Homozygous for CYP2J2*7 (wild type for the other SNPs)

EXCLUSION CRITERIA:

1. Current pregnancy or lactation, as medications used during the bronchoscopy can be excreted in the breast milk of lactating mothers
2. Current smoker or significant second-hand smoke exposure (defined by urine cotinine >200 ng/mL at screening)
3. Post-bronchodilator FEV1 < 70% of predicted
4. For asthmatics, any indication of moderate or severe asthma such as:

   * Physician-directed emergency treatment for an asthma exacerbation within the preceding 12 months
   * Any use of systemic steroid therapy during the last year or continuous use of inhaled steroids over a period of 1 month or longer during the past 6 months
   * Regular use of cromolyn (except for prophylaxis of exercise induced bronchospasm) or any use of leukotriene inhibitors (Montelukast or Zafirlukast) within the past month
   * Symptoms including:

     * Night-time symptoms of cough or wheeze greater than 1x/week
     * Exacerbations of asthma more than 2x/week
     * Daily requirement for albuterol due to asthma symptoms (cough, wheeze, chest tightness)
5. Bleeding disorders or regular use of aspirin or other non-steroidal anti-inflammatory drugs (which inhibit platelet function) or other drugs that prolong bleeding time such as warfarin, heparin or derivatives, or clopidogrel and related ADP inhibitors
6. Sickle cell disease or GP6 deficiency
7. Facial deformity or major facial surgery
8. Asthma exacerbation or respiratory infection 4 weeks prior to study visit
9. Allergy or history of adverse reactions to lidocaine, midazolam, or fentanyl
10. Vital signs (temperature, blood pressure, pulse rate) that are outside of the established CRU limits
11. Body weight <50 kg (<110 lbs)
12. The following abnormal clinical laboratory values (obtained during Visit 1 assessment):

    * Platelet count <100,000 per L
    * White blood cells count <3000 per L
    * Absolute neutrophil count <1000 per L
    * Hematocrit <35% for both female and male
    * PT/INR and PTT based on reference laboratory established reference ranges
    * Serum creatinine >1.4 mg/dL
13. Any condition that, in the investigator's opinion, places the participant at undue risk for complications associated with required study procedures.
14. Use of the medication colchicine (commonly used to treat gout attacks) in the past 2 weeks.

Volunteers meeting any of the below temporary exclusions may enroll in the study, but may not

undergo the bronchoscopy procedure within the time frames specified for each below temporary exclusion. If any of the following conditions are met, the bronchoscopy will be rescheduled such that none of these temporary exclusions apply:

Temp. EXCL 1. An asthma exacerbation requiring increased asthma medications for more than 1 day (and other than exercise-induced asthma) within 1 month of bronchoscopy

Temp. EXCL 2. Viral upper respiratory tract infection or any acute infection requiring antibiotics within 4 weeks of bronchoscopy

Temp. EXCL 3. Use of anti-inflammatory medications (including over-the-counter preparations) during the 48 hours prior to the bronchoscopy and aspirin during the 14 days prior to bronchoscopy.

Temp. EXCL 4. Any food or fluids for 8 hours prior to the bronchoscopy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2019-12-18 (Actual); Study Completion 2023-09-21 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure will evaluate macrophage phagocytosis of fluorescein isothiocyanate (FITC)-labeled beads and bacteria (Streptococcus pneumoniae) in an ex vivo assay, comparing alveolar macrophages from groups of individuals with and ... | Cross-sectional
  The primary outcome measure will evaluate macrophage phagocytosis of fluorescein isothiocyanate (FITC)-labeled beads and bacteria (Streptococcus pneumoniae) in an ex vivo assay, comparing alveolar macrophages from groups of individuals with and without EPHX2 and CYP2J2 polymorphisms of interest.

CONTACTS AND LOCATIONS:
Overall Officials: Darryl C Zeldin, M.D., Principal Investigator — National Institute of Environmental Health Sciences (NIEHS)
Locations (1):
- NIEHS, Research Triangle Park, Research Triangle Park, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided
It isn t known yet if there will be a plan to make IPD available

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2016-E-0096.html